CLINICAL TRIAL: NCT03381313
Title: Improving Word Repetition Training Using Classical Conditioning With a Computer Based Telemedicine Approach: Evidence From a Study on 12 Person With Chronic Aphasia.
Brief Title: Classical Conditioning Training for Aphasia. A Telemedicine Approach.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Giovanni Augusto Carlesimo, Principal Investigator, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: 12 patients suffering from pure anomia in the chronic stage of the disease underwent a word repetition training with a computerized telemedicine protocol. Each patient trained two word sets, one in a conditioned and the other in a non-conditioned training modality; a third non trained set served as control.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anomic Patients (Experimental): Pure Anomic Patients underwent to conditioned word repetition training or traditional one.
  Interventions: Behavioral: Conditioned word repetition training

INTERVENTIONS:
Behavioral: Conditioned word repetition training — In the classical conditioning training the onset of the visual stimulus preceded that of the auditory stimulus with a short onset asynchrony, and both stimuli co-terminated. By contrast, in the training without conditioning the auditory stimulus was administered first and the visual stimulus appeared short after the off-set of the auditory one.

SUMMARY:
This study aimed at investigating the suitability of a classical conditioning for the treatment of anomic disorder. In this study 12 patients suffering from pure anomia in the chronic stage of the disease underwent a word repetition training with a computerized telemedicine protocol. Each patient trained two word sets, one in a conditioned and the other in a non-conditioned training modality; a third non trained set served as control set.

DETAILED DESCRIPTION:
In this study, a computer based word repetition protocol was administered at the distance to 12 pure anomic patients in the chronic stage of the disease. The to be repeated words were presented alongside the corresponding pictures. The timing of word and picture presentation was manipulated in order to investigate the suitability of classical conditioning to reteach the association between pictures and their names. Data were analyzed at the group and at the single subject level with the aim of establishing the relative efficacy of the conditioned and non-conditioned word-repetition modality and the cognitive features predicting therapy success. In keeping with preliminary results obtained on a single case study, conditioning turned out to improve therapy gain at the group level. Moreover, hints were found suggesting less generalization to untreated words in conditioned compared to non-conditioned training. Non-word repetition skills was the only feature in the participants cognitive profile which was reliably linked to the therapy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Aphasic patients with word finding difficulty
* Must be able to repeat single words

Exclusion Criteria:

* Severe cognitive impairment
* Impaired single word comprehension

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Training effect in the treated word set | immediately before and immediately after the training protocol (duration of the training protocol: 6 weeks)
  Differences between accuracy pre and post in the treated word set

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni A Carlesimo, MD, Principal Investigator — I.C.C.S Fondazione Santa Lucia

IPD SHARING:
Plan to Share IPD: No